CLINICAL TRIAL: NCT03053882
Title: Comparative Study of the Effects of Green Tea and Peppermint Herbal Mouthwash on Halitosis.
Brief Title: Efficacy of Peppermint and Green Tea in Malodor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mahin Bakhshi, Associate Professor of Oral Medicine, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: SBMU
Record Dates: First submitted 2017-02-04; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Bad Breath
Keywords: mouth wash , green tea , peppermint , bad breath
MeSH Terms: conditions — Halitosis | interventions — Mouthwashes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- green tea and peppermint (Active Comparator)
  Interventions: Other: mouthwash
- peppermint and green tea (Active Comparator)
  Interventions: Other: mouthwash

INTERVENTIONS:
Other: mouthwash — mouthwash containing herbal peppermint or green tea

SUMMARY:
Background:

Herbal remedies can have the role of prevention and control of bad breath Since in the previous studies, therapeutic and antibacterial effect of green tea and peppermint had been proven .we studied and compared the effects of green tea and peppermint mouthwashes on halitosis.

Materials and Methods:

This single-blind clinical trial study with cross over design total of 88 volunteer dental students who complained bad breath and had organoleptic score (>= 2) and higher average test scores were enrolled. The students were divided randomly into two groups Green Tea - Peppermint were assigned. Organoleptic test in the baseline, on the 7 day, 14 and 21 measured after rinsing the mouthwashes .As well as the satisfaction of both plants on the last day was considered. Data analysis was performed using tests; Wilcoxon signed rank test, Mann Whithney u, GEE (Generalized Estimating Equation -ordinal logistic regression).

ELIGIBILITY:
Inclusion Criteria:

organoleptic number equal to or higher 2 no foods (garlic and onion) 48 hours before organoleptic test

Exclusion Criteria:

systemic disease

* use of antibiotics during study use of other mouthwash during study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
evaluation of changes in organoleptic score | baseline,7 days,14 days,21 days
  0-5 organoleptic scale

SECONDARY OUTCOMES:
satisfaction of patients | 21 days
  questionnaire